CLINICAL TRIAL: NCT04545450
Title: A Randomized Double-blind Placebo-controlled Pilot Trial on the Effects of Testosterone Undecanoate Plus Dutasteride or Placebo on Muscle Strength, Body Composition and Metabolic Profile in Transmen
Brief Title: Effects of Testosterone Plus Dutasteride or Placebo on Muscle Strength, Body Composition and Metabolism in Transmen
Acronym: DUTMUSCLE-20
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unita Complessa di Ostetricia e Ginecologia (Other)
Responsible Party: Principal Investigator, maria cristina meriggiola, Principal Investigator, Unita Complessa di Ostetricia e Ginecologia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUTMUSCLE-20
Record Dates: First submitted 2020-08-10; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Transgenderism; Hypogonadism
Keywords: Muscle strenght; Testosterone; Dutasteride; dihydrotestosterone; 5a-reductase inhibitor
MeSH Terms: conditions — Transsexualism; Hypogonadism | interventions — Dutasteride; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the research pharmacist was aware of the randomization results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testosterone Undecanoate plus dutasteride (Active Comparator): Testosterone Undecanoate (TU) 1000 mg i.m. at weeks zero, six, 18, 30, 42 + dutasteride 5 mg/day
  Interventions: Drug: dutasteride 5 mg/day; Drug: Testosterone Undecanoate
- Testosterone Undecanoate plus placebo (Placebo Comparator): Testosterone Undecanoate (TU) 1000 mg i.m. at weeks zero, six, 18, 30, 42 + a daily oral placebo pill
  Interventions: Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: dutasteride 5 mg/day — Administration of a placebo pill or dutasteride 5 mg pill daily in addition to intramuscolar testosterone undecanoate
  Arms: Testosterone Undecanoate plus dutasteride
Drug: Testosterone Undecanoate — Administration of a placebo pill or dutasteride 5 mg pill daily in addition to intramuscolar testosterone undecanoate

SUMMARY:
To compare the effects on body composition and muscle strengthof 54-weeks treatment with of testosterone undecanoate combined with placebo or with the 5a-reductase inhibitor dutasteride

DETAILED DESCRIPTION:
Transmen who have undergone gender-affirming surgery require long-lasting treatments with androgens to maintain male phenotypic characteristics and to preserve their health. In this population the effects on muscle and the relative role of testosterone and its metabolite dihydrotestosterone (DHT) on the skeletal muscle are still largely unknown.

In this pilot study, we evaluated the effects of testosterone and DHT on muscle strength, body composition, metabolism. Also cutaneous androgenic effects such as acne and androgenetic alopecia were evaluated.

DESIGN

For this purpose, in this randomized, double-blind placebo-controlled pilot trial we treated variectomized transmen for 54 weeks with:

* Testosterone Undecanoate (TU) 1000 mg i.m. at weeks zero, six, 18, 30, 42 + a daily oral placebo pill (TU+PL)
* TU 1000 mg i.m. at weeks zero, six, 18, 30, 42 + dutasteride 5 mg/day (TU+DUT).

Prospective, phase III, randomized study design was used.

Subjects were seen every 12 weeks for safety monitoring that included evaluation of hematocrit, transaminases, alkaline phosphatases and bilirubin, creatinine, urea and serum electrolyte as potassium and sodium.

Baseline and week-54 evaluations included the following measurements:

blood drawings for measurements of: hormonal profile (serum testosterone, estradiol, luteinizing hormone and follicle-stimulating hormone, prolactin, sex hormone binding globulin, and thyroid stimulating hormone), haematocrit (Ht) and haemoglobin (Hb), glucidic and lipidic profile (fasting glucose, fasting insulin, total cholesterol, high- and low-density lipoproteins, and triglycerides), hepatic function (aspartate and alanine aminotransferases) and bone related markers (osteocalcin, parathyroid hormone, bone alkaline phosphatase and 25-hydroxyvitamin, 24h urinary excretion of calcium, potassium, magnesium and creatinine).

anthropometry: weight, measures DEXA for bone mass determination and body composition Isokinetic knee extension and flexion peak torque (PT-IKE and PT-IKF) Handgrip strength evalutation of the psychological profile with the brief Profile of Mood State (POMS) sexual life satisfaction evalutation with a Visual Analogue General Satisfaction Scale (VAS) physical examination: inspection of external genitalia (clitorides) and a visit to detect appearance of acne and gynecomastia

During the treatment phase all injections will be administered by the investigator or co-investigators for the entire study. Fasting (10 hours) blood samples will be taken (immediately before giving the injections) every time subjects come for injections (week 0, 6, 18, 30 and 42) and at the end of the treatment phase.

In the sexual and behavior questionnaire the subjects will judge their sexual activity and behavior in the period between visits. The subjects have the possibility to making additional comments about important events and disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Healthy transmen
* Previous bilateral gonadectomy during sex reassigning surgery
* Body Mass Index (BMI) between 20 and 29 kg/m²; (body weight in kilograms divided by body height in meters squared)
* Clinical examination without pathological findings relevant to the study
* No concomitant use of drugs known to affect the hypothalamic-pituitary-ovarian axis
* Written Consent Form
* High probability of a good compliance and termination of the study

Exclusion Criteria:

* Participation in another clinical trial within the 30 days preceding the first administration
* Simultaneous participation in another clinical trial
* Subjects institutionalized or imprisoned by order of the court
* Subject who compete in sports
* Subjects reporting desire to perform regular physical exercises for the duration of the study
* Serious organic or psychic disease suspected from history and/or clinical examination
* Diseases (especially tumors) that might represent an actual contraindication for testosterone
* Past or present history of thrombotic or embolic diseases
* Arterial hypertension
* Diabetes mellitus
* Acute or chronic hepatic diseases
* Manifest renal diseases with renal dysfunction
* Severe internal diseases
* Biochemical and/or hematological laboratory values beyond normal ranges unless the Investigator confirms that the deviations are of no clinical relevance
* Any indication of chronic use of drugs, alcohol, opiates or recreational drugs
* Use of any drug known to affect biotransformation of testosterone and/or progestin, e.g. chlorcycline, phenobarbital, phenylbutazone, aminophenazone within the 30 days preceding the first administration of the test medication and during the study
* Use of oral anticoagulatory drugs within the 30 days preceding the first administration of the test medication and during the study
* Any oral or transdermal hormone medication within the 12 weeks preceding the first administration and during the study
* Probability of poor compliance and termination of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11-04 (Actual); Primary Completion 2009-07-30 (Actual); Study Completion 2010-10-15 (Actual)

PRIMARY OUTCOMES:
Change in isokinetic knee extension and flexion peak torque (PT-IKE and PT-IKF) | At baseline and after 54 weeks of treatment
  Isokinetic peak torques were determined using isokinetic dynamometry (Biodex System 4 Pro, Medical Systems, Shirley, NY) at all four time points.
Change in handgrip strength | At baseline and after 54 weeks of treatment
  Three trials of three sets of maximal isometric handgrip on a mechanical dynamometer (model Grip-A, Takei Physical Fitness Test TKK 5001, Japan), alternately with the dominant and non-dominant hand, with a three minute rest between each trial
Change in body composition | At baseline and after 54 weeks of treatment
  Dual-energy X-ray absorptiometry was performed using the Hologic 49159 densitometer and standard QDR body composition software (Model QDR4500W, Software Level 11.2, Hologic Spine; Hologic, Bedford, MA) for the measurement of body fat and lean mass
Change in bone mineral density | At baseline and after 54 weeks of treatment
  Dual-energy X-ray absorptiometry was performed using the Hologic 49159 densitometer and standard QDR body composition software (Model QDR4500W, Software Level 11.2, Hologic Spine; Hologic, Bedford, MA) for the evaluation of bone mineral density at lumbar and femoral site
Change in anthropometric assessment: BMI | At baseline and after 54 weeks of treatment
  weight, stature will be combined to report the BMI (kg/m^2)
Change in anthropometric assessment: waist-to-hip ratio | At baseline and after 54 weeks of treatment
  Waist and hip circumferences will be combined to report the waist-to-hip ratio (WHR)

SECONDARY OUTCOMES:
Change in psychological profile with the brief Profile of Mood State (POMS) | At baseline and after 54 weeks of treatment
  The POMS is a self-reporting questionnaire consisting of 30 items in six categories: tension-anxiety, depression, anger-hostility, vigor, fatigue and confusion, which are scored from 1-4 according to severity
Change in the satisfaction with their sexual life | At baseline and after 54 weeks of treatment
  using a Visual Analogue General Satisfaction Scale (VAS). A VAS for satisfaction is a horizontal line of 10-cm long. At the start and finish there are two descriptors representing extremes of satisfaction (i.e. no satisfaction and extreme satisfaction). Subjects respond to the question 'Are you satisfied with your sexual life now?' and rate their satisfaction by making a vertical mark on the 100-mm line. The measurement in millimeters is converted to the same number of points ranging from zero to 10 points.
Change in in the bone metabolism: osteocalcin | At baseline and after 54 weeks of treatment
  Evaluation of serum osteocalcin (OC) change
Change in in the bone metabolism: parathyroid hormone | At baseline and after 54 weeks of treatment
  Evaluation of serum parathyroid hormone (PTH) changes
Change in in the bone metabolism: bone alkaline phosphatase | At baseline and after 54 weeks of treatment
  Evaluation of serum bone alkaline phosphatase (BAP) changes
Change in in the bone metabolism: urinary excretion of electrolites | At baseline and after 54 weeks of treatment
  Changes in the 24h urinary excretion of electrolites
Change in in the insulin resistance | At baseline and after 54 weeks of treatment
  Change in the HOMA-IR (Homeostatic Model Assessment for Insulin Resistance)
Change in the lipid profile | At baseline and after 54 weeks of treatment
  Changes in cholesterol (Tot Chol and high- and low-density lipoproteins) levels
Change in the lipid profile | At baseline and after 54 weeks of treatment
  Changes in triglycerides levels